CLINICAL TRIAL: NCT04343586
Title: Development & Preliminary Clinical Validation Blue Light Phototherapy Systems for T-Cell
Brief Title: Blue Light Phototherapy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Northwestern University (Other)
Collaborators: T-Cellerate LLC (Industry)
Responsible Party: Principal Investigator, Shuai (Steve) Xu, Principal Investigator, Northwestern University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STU00210472
Record Dates: First submitted 2020-01-24; First posted 2020-04-13 (Actual); Results first posted 2023-03-17 (Actual); Last update posted 2023-03-17 (Actual); Status verified 2023-02

CONDITIONS: Grover's Disease; Psoriasis Vulgaris
MeSH Terms: conditions — Grover's disease | interventions — Phototherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Adult treatment arm (Experimental): Adults enrolled in the study will receive treatment (blue light phototherapy) on one area of their body affected by psoriasis or Grover's disease. The treatment area (restricted by size of the device) will be compared to untreated areas affected by disease on the same patient.
  Interventions: Device: Blue light phototherapy

INTERVENTIONS:
Device: Blue light phototherapy — Phototherapy- Wavelength: 417±15 nm
  Other Names: DusaPharma Blu-U model 4170

SUMMARY:
This study will use Blue-light Photo-therapy to treat patients with psoriasis vulgaris and Grover's Disease.

ELIGIBILITY:
Inclusion Criteria:

1. Patient's aged 18-89 at time of enrollment
2. Previous diagnosis of psoriasis vulgaris or Grover's disease

Exclusion Criteria:

1. All Groups: Subjects who are younger than 18 years of age or older than 90 years of age
2. Patients who have received topical or systemic treatment within the prior 2 weeks of planned phototherapy
3. Patients prescribed any of the following drugs for issues not related to their psoriasis or Grover's disease

   * topical steroids
   * calcineurin inhibitors
   * methotrexate
   * retinoids
   * biologic agents
4. Unable to schedule phototherapy sessions
5. We will not recruit the following populations: adults unable to consent, individuals who are not yet adults (infants, children, teenagers), pregnant women, prisoners and other vulnerable populations.

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2020-09-01 (Actual); Primary Completion 2021-12-20 (Actual); Study Completion 2022-09-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Shuai Xu, Principal Investigator — Northwestern University
Locations (1):
- Northwestern University Department of Dermatology, Chicago, Illinois, United States

REFERENCES:
- [Derived] Olagbenro M, Ravi S, Myers D, Lin D, Woodburn W, Walter JR, Xu S. Assessment of Blue Light Phototherapy for Grover Disease: A Nonrandomized Controlled Trial. JAMA Dermatol. 2023 Jan 1;159(1):102-104. doi: 10.1001/jamadermatol.2022.4491. PMID 36449285

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Adult Treatment Arm
Started | 11
Completed | 10
Not Completed | 1

BASELINE CHARACTERISTICS:
Arm/Group | Adult Treatment Arm
Number analyzed (Participants) | 11
Age, Continuous [Mean (Standard Deviation); unit: years] | 63 (14)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 9
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 11

OUTCOME MEASURES:

1. Primary Outcome: Efficacy of Blue Light Therapy for Patients With Grover's Disease
Description: Demonstrate preliminary skin efficacy as measured by lesion count
Time Frame: Time Frame: 5 weeks
Measure: Mean (95% Confidence Interval); unit: lesion count
Arm/Group | Adult Treatment Arm
Number analyzed (Participants) | 10
lesion count
  Baseline | 27 [9.2 to 45.6]
  End of Treatment | 6 [2.5 to 8.7]

2. Primary Outcome: Assess User Experience With the Dermatology Life Quality Index (DLQI) Pre and Post-treatment.
Description: The DLQI is a questionnaire with 10 questions. The maximum score is 30 and minimum is 0. The higher the score, the more quality of life is impaired.
Time Frame: Time Frame: 5 weeks
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Adult Treatment Arm
Number analyzed (Participants) | 10
score on a scale
  Baseline | 4.3 [1.3 to 7.4]
  End of Treatment | 2.3 [1.3 to 3.4]

ADVERSE EVENTS:
Time Frame: 5 weeks
Arm/Group | Adult Treatment Arm
All-Cause Mortality (participants affected / at risk) | 0/11
Serious Adverse Events (participants affected / at risk) | 0/11
Other Adverse Events (participants affected / at risk) | 0/11

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-07-26): https://cdn.clinicaltrials.gov/large-docs/86/NCT04343586/Prot_SAP_000.pdf
  • Informed Consent Form (2021-08-02): https://cdn.clinicaltrials.gov/large-docs/86/NCT04343586/ICF_001.pdf